CLINICAL TRIAL: NCT06423456
Title: A New Alternative for Postoperative Pain Control Following Hysteroscopy;Preoperative Intravenous Lidocaine
Brief Title: Postoperative Pain Control Following Hysteroscopy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Afyonkarahisar Health Sciences University (Other)
Responsible Party: Principal Investigator, Betül Ahat, Assistant Doctor, Afyonkarahisar Health Sciences University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: AFSU-OBGYN-BA-01
Record Dates: First submitted 2024-05-16; First posted 2024-05-21 (Actual); Results first posted 2025-07-23 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2025-07

CONDITIONS: Postoperative Pain; Postoperative Nausea; Analgesia
Keywords: hysteroscopy; intraoperative lidocaine; postoperative pain; postoperative nausea
MeSH Terms: conditions — Pain, Postoperative; Postoperative Nausea and Vomiting; Agnosia | interventions — Sodium Chloride

STUDY DESIGN:
Intervention Model Description: Intraoperative lidocaine infusion is a frequently preferred method in surgical procedures due to its reducing the need for opioids, providing better postoperative pain control, reducing postoperative nausea and vomiting and increasing rapid recovery. Our aim in this study is to show the effect of intraoperative lidocaine infusion on reducing complications such as pain, nausea, vomiting, and the need for opioid analgesia that occur after hysteroscopy operations, which are often performed in gynecology clinics.
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Research group (Active Comparator): During the procedure, intravenous lidocaine of 0.15 ml/kg 1% will be administered intraoperatively before general anesthesia and infusion of lidocaine of 1%(at a dose of 0.2 ml/kg/hour) will be performed during the procedure.
  Interventions: Drug: Lidocaine IV
- Control group (Placebo Comparator): In the control group, 0.9% saline solution will be used instead of lidocaine.
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: Lidocaine IV — Pain measurement will be performed using a visual analog scale (VAS) for postoperative pain after the operation. At the same time, patients' intraoperative analgesic use, postoperative nausea-vomiting and antiemetic use will be recorded.
  Other Names: lidocaine HCl 2%
  Arms: Research group
Drug: Saline — Pain measurement will be performed using a visual analog scale (VAS) for postoperative pain after the operation. At the same time, patients' intraoperative analgesic use, postoperative nausea-vomiting and antiemetic use will be recorded.
  Other Names: 0.09% Saline
  Arms: Control group

SUMMARY:
Intraoperative lidocaine infusion is a frequently preferred method in surgical procedures due to its reducing the need for opioids, providing better postoperative pain control, reducing postoperative nausea and vomiting and increasing rapid recovery. Our aim in this study is to show the effect of intraoperative lidocaine infusion on reducing complications such as pain, nausea, vomiting, and the need for opioid analgesia that occur after hysteroscopy operations, which are often performed in gynecology clinics.

DETAILED DESCRIPTION:
Hysteroscopy abnormal uterine bleeding, infertility, endometrial pathologies, uterine fibroids,it is a method that is often used in the diagnosis and treatment of pathologies such as intrauterine synechia.

Hysteroscopy; observation of the inner layer of the uterus with a special optical instrument with a cold light source and it is the process of making intrauterine interventions using small hand tools. General anesthesia or with intrauterine fluid after dilating the cervix under regional (epidural/peridural) anesthesia it is filled and a thin telescope-like optical device (hysteroscope) is transmitted into the uterus. This way the uterine cavity is observed. Hysteroscopy is used for diagnostic purposes as well as for therapeutic purposes it can be applied.

General Anesthesia (GA) is often the preferred method for operative hysteroscopy.Intraoperative lidocaine infusion reduces the need for opioids, postoperative pain control is better due to the fact that it reduces postoperative nausea, vomiting and increases rapid recovery, which is often preferred in surgical procedures. 150 patients who are scheduled to undergo hysteroscopy will be included in the study. Hysteroscopy the patients to be applied will be divided into two groups as research and control groups. To both groups 75 patients will be included each. General anesthesia during the procedure for patients in the research arm intravenous lidocaine of 0.15 ml/kg 1% will be administered intraoperatively before and during the procedure a 1% lidocaine infusion(at a dose of 0.2 ml/kg/hour) will be performed. In the control group, if 0.9% saline solution will be used instead of lidocaine.

Pain measurement using visual analog scale (VAS) for postoperative pain after surgery will be done. At the same time, intraoperative analgesic use of patients, postoperative nausea-vomiting and antiemetic uses will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Female patients with ASA I-II according to the American Society of Anesthesiologists (ASA) classification who are scheduled for elective hysteroscopy with indications such as
* abnormal uterine bleeding
* endometrial polyp
* submucosal myoma
* foreign body in the endometrial cavity
* infertility
* intrauterine synechia

Exclusion Criteria:

* Patients under the age of 18
* Who are allergic to lidocaine addicted to opioids or NSAIDs
* Patients with chronic pain
* Patients with severe systemic disease
* Patients who do not approve

Ages: 19 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 150 (Actual)
Dates: Start 2024-03-01 (Actual); Primary Completion 2025-02-23 (Actual); Study Completion 2025-02-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Betul Ahat, Principal Investigator — Afyonkarahisar University of Health Science, school of medicine; Tuba Berra Sarıtaş, Study Chair — Afyonkarahisar University of Health Science, school of medicine; Rıza Dur, Study Director — Afyonkarahisar University of Health Science, school of medicine
Locations (1):
- Afyonkarahisar University of Health Science, school of medicine, hospital, Merkez, Afyonkarahi̇sar, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Research Group | Control Group
Started | 75 | 75
Completed | 75 | 75
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: patients who are scheduled to undergo hysteroscopy will be included in the study. All participants were included in the study
Groups:
- Total: Total of all reporting groups
Arm/Group | Research Group | Control Group | Total
Number analyzed (Participants) | 75 | 75 | 150
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 75 | 75 | 150
  >=65 years | 0 | 0 | 0
Age, Continuous [Median (Standard Deviation); unit: years] | 39.96 (7.87) | 41.95 (8.83) | 40.6 (7.91)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 75 | 75 | 150
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 75 | 75 | 150
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Turkey | 75 | 75 | 150

OUTCOME MEASURES:

1. Primary Outcome: Visual Analog Scale (VAS)
Description: After the hysteroscopy procedure is completed, in the postoperative anesthesia care room, postoperative, 30. and 60. in minutes, 4. per hour and 24. pain measurement will be performed for patients per hour using a visual analog scale (VAS) for postoperative pain. In this scale, patients' pain between 0-10 (0=no pain, 10=very severe pain) will be questioned. Dec. The doctor who performed the measurement will not know which drug infusion was made. NSAIDs will be administered to patients with a VAS score > 4. Opioid analgesics will be administered to patients whose pain does not go away. At the same time, patients' intraoperative analgesic use, postoperative nausea-vomiting and antiemetic use will be recorded.
Time Frame: 24 hours
Measure: Median (Standard Deviation); unit: score on a scale
Arm/Group | Research Group | Control Group
Number analyzed (Participants) | 75 | 75
score on a scale
  postoperative 30th minute | 2.49 (1.61) | 4.44 (1.88)
  postoperatice 60th minute | 1.23 (1.07) | 2.40 (1.58)
  postoperative 4.hour | 0.61 (0.28) | 1.09 (1.08)
  postoperative 24.hour | 0.20 (0.04) | 0.63 (0.36)

ADVERSE EVENTS:
Time Frame: ADVERSE EVENT DATA WERE COLLECTED FOR 1 WEEK AFTER THE PROCEDURE
Arm/Group | Research Group | Control Group
All-Cause Mortality (participants affected / at risk) | 0/75 | 0/75
Serious Adverse Events (participants affected / at risk) | 0/75 | 0/75
Other Adverse Events (participants affected / at risk) | 0/75 | 0/75

LIMITATIONS AND CAVEATS:
Comprise relatively small cohort size, lack of preoperative VAS score, heterogeneity related with the type of hysteroscopy and operative findings.That the hysteroscopy procedure was not performed by the same surgeon. The inability to measure plasma lidocaine level in this study can be identified. However, since no adverse effects occurred due to IV lidocaine treatment in the postoperative period, it is thought that the toxic dose was not reached in any patient.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (3):
  • Study Protocol (2024-11-07): https://cdn.clinicaltrials.gov/large-docs/56/NCT06423456/Prot_000.pdf
  • Statistical Analysis Plan (2024-12-24): https://cdn.clinicaltrials.gov/large-docs/56/NCT06423456/SAP_001.pdf
  • Informed Consent Form (2024-02-26): https://cdn.clinicaltrials.gov/large-docs/56/NCT06423456/ICF_002.pdf